CLINICAL TRIAL: NCT02127905
Title: A Study of Total Body Irradiation, Cyclophosphamide and Fludarabine Followed by Alternated Donor Hematopoietic Cell Transplantation in Patients With Fanconi Anemia
Brief Title: Unrelated HSCT in Patients With Fanconi Anemia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to non-enrollment of subjects due to rarity of disease.
Sponsor: Neena Kapoor, M.D. (Other)
Responsible Party: Sponsor-Investigator, Neena Kapoor, M.D., Professor of Pediatrics, Keck School of Medicine; Division Head, Division of Research Immunology/BMT, Children's Hospital Los Angeles
Organization: Children's Hospital Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI-10-00176
Record Dates: First submitted 2012-10-19; First posted 2014-05-01 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Fanconi Anemia
Keywords: Fanconi Anemia; compassionate treatment; BMT; HSCT; unrelated; bone marrow transplantation; PBSC; peripheral blood; CD34+
MeSH Terms: conditions — Fanconi Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CD34+ selected cells (Other): use of unrelated bone marrow or peripheral blood for hematopoietic stem cell transplantation with CD34+ selected cells
  Interventions: Biological: CD34+ selected cells

INTERVENTIONS:
Biological: CD34+ selected cells — Compassionate treatment of Fanconi Anemia patients with unrelated bone marrow or peripheral blood HSCT followed by the infusion of CD34+ selected cells using CliniMACS
  Other Names: CD34+ selected cells using CliniMACS

SUMMARY:
The protocol is designed for the compassionate treatment of patients with Fanconi Anemia who do not have an HLA-matched sibling donor. The purpose of this study is to determine the likelihood of engraftment in Fanconi Anemia patients using total body irradiation (TBI), cyclophosphamide (CY), fludarabine (FLU) and antithymocyte globulin (ATG) followed by an unrelated donor hematopoietic cell transplant with T-cell depletion using the CliniMACS device.

DETAILED DESCRIPTION:
The major obstacle to successful alternate donor HCT for patients with Fanconi Anemia is graft failure. While T-cell depletion decreases the incidence of aGVHD, its effect on improving long term survival is unproven. To potentially improve engraftment rate, we have chosen a relatively new immunosuppressive agent, fludarabine (FLU), FLU is an antineoplastic agent that has been shown to be an effective immunosuppressive agen in BMT conditioning therapy. The addition of FLU to the commonly used preparative regimen of CY and TBU in Fanconi Anemia patients may improve engraftment rates.

Based on all presented data and its outcome, hematopoietic stem cell transplantation with the use of total body irradiation (450 cGy), cyclophosphamide (10 mg/kg IV) and fludarabine (35 mg/m2 IV) as preparative cytoreductive therapy has become the standard treatment for the hematologic manifestations of Fanconi Anemia at CHLA. However, the use of Isolex 300i will be replaced by CliniMACS in processing T-cell depletion.

The CliniMACS CD34 Reagent System is an investigational medical device that has not yet been approved by the FDA. This device is used in vitro to select and enrich specific cell populations. When using the CliniMACS CD34 Reagent, the system selects CD34+ cells from heterogenous hematological cell populations for transplantation in cases where this is clinically indicated. Based on the gathered data, CliniMACS has not been a contributing factor in the toxicity of patients, although may have a potential of eliciting "antibody" reactions in some patients, the process has been of significant life-saving benefit as compared to the potential risks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > 2 months and < 21 years of age with a diagnosis of Fanconi anemia.
* Patients must have an HLA-A, B, DRB1 identical or 1 antigen mismatched related (non-sibling) or unrelated donor. Patients and donors will be typed for HLA-A and B using serological or molecular techniques and for DRB1 using high resolution molecular typing. (Patients with a 2 antigen mismatched related donor will be eligible for the protocol but evaluated separately).
* Patients with FA must have high risk genotype or aplastic anemia (AA) or myelodysplastic syndrome without excess blasts.
* Aplastic anemia is defined as having at least one of the following:

  1. platelet count <20 x 109/L
  2. ANC <5 x 108/L
  3. Hgb <8 g/dL with at least one of the following:

  <!-- -->

  1. transfusion dependence
  2. supportive care toxicity
* Myelodysplastic syndrome with multilineage dysplasia with or without chromosomal anomalies.
* High risk genotype (e.g. IVS-4 or exon 14 FANCC mutations)
* Adequate major organ function including:
* Cardiac: ejection fraction >45%
* Renal: creatinine clearance >40 mL/min.
* Hepatic: no clinical evidence of hepatic failure (e.g. coagulopathy, ascites)
* Karnofsky performance status >70% or Lansky >50%
* Women of child bearing age must be using adequate birth control and have a negative pregnancy test.

Exclusion Criteria:

* Available HLA-genotypically identical related donor.
* The harvested marrow (prior to TCD) should contain a minimum of 2.5 x 108 nucleated cells/kg recipient body weight with a goal of >5.0 x 108 nucleated cells/kg recipient body weight.
* Positive lymphocytotoxic crossmatch against donor (T cells and B cells)
* History of gram negative sepsis or systemic fungal infection (proven or suspected based on radiographic studies).
* Myelodysplastic syndrome with excess blasts or leukemia.
* Active CNS leukemia at time of HCT.
* Malignant solid tumor (e.g. squamous cell carcinoma of the head/neck/cervix) within 2 years of HCT.
* Pregnant or lactating female.
* Prior radiation therapy preventing use of TBI 450 cGy.

Ages: 8 Weeks to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03 (Estimated); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Event free survival post stem cell transplant | 5 years
  Patients who are alive at 5 years post transplants with assessments at 30, 60, 90, 180 and yearly up to 5 years

SECONDARY OUTCOMES:
Peripheral blood CBC counts for engraftment evaluation | 3 years
  Normalization of Hemoglobin, platelets and neutrophil count
Chimerism assay for engraftment evaluation | 3 years
  Assessment of chimerism by FISH or STR on peripheral blood and bone marrow
Graft Versus Host Disease (GVHD) surveillance after HSCT | 3 years
  GHVD disease surveilance done by clinical evaluation, to include history, physical examination, specifically for rash, jaundice, liver dysfunction, nausea and vomiting, diarrhea and failure to thrive

CONTACTS AND LOCATIONS:
Overall Officials: Neena Kapoor, M.D., Principal Investigator — Children's Hospital Los Angeles, University of Southern California
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Procedure as well as de-identified data is reported to CIBMTR and is available to other researchers.
Supporting Information: Study Protocol, CSR
Time Frame: End of subject enrollment and following 2 year subject follow-up
Access Criteria: Researchers/Investigators interested in severe combined immune deficiency disease treatment and outcomes.